CLINICAL TRIAL: NCT02643589
Title: Dose Study of Antithymocyteglobulin in Haploidentical Hematopoietic Stem Cell Transplantation for Acute Graft-versus-host Disease Prophylaxis
Brief Title: Dose Study of Antithymocyteglobulin in Haploidentical Allogeneic Stem Cell Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Peking University People's Hospital (Other); Central South University Xiangya Hospital (Unknown); Fujian Medical University (Other)
Responsible Party: Principal Investigator, Qifa Liu, Professor, Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NFEC-201304-K1(02)
Record Dates: First submitted 2015-12-29; First posted 2015-12-31 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: Hematopoietic Stem Cell Transplantation
Keywords: haploidentical hematopoietic Stem Cell Transplantation Antithymocyte globulin; acute graft-versus-host disease; antithymocyte globulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ATG 7.5mg/kg (Experimental): ATG 7.5mg/kg group refers to treatment with ATG in the total dose of 7.5mg/kg.
  Interventions: Drug: ATG
- ATG 10mg/kg (Active Comparator): ATG 10mg/kg group refers to treatment with ATG in the total dose of 10mg/kg.
  Interventions: Drug: ATG

INTERVENTIONS:
Drug: ATG — ATG will be intravenously infused via a central venous catheter in 3 or 4 days, from day -4 or -3 until day 0. The other conditioning drugs administered before transplantation include cytosine arabinoside (Ara-C), busulfan (Bu),cyclophosphamide (Cy), Semustine(Me-CCNU), and ATG. All transplant recipients will receive cyclosporine A (CsA), mycophenolate mofetil(MMF), and short-term methotrexate for aGVHD prevention.

SUMMARY:
The purpose of this study is to compare the incidences of GVHD in haploidentical hematopoietic stem cell transplant recipients receiving different dose of antithymocyte globulin (ATG) for acute graft-versus-host disease(aGVHD) prophylaxis. The investigators' first objective was to investigate the optimal dose of ATG for aGVHD.

DETAILED DESCRIPTION:
Graft-versus-host diseases (GVHD) remains a major cause of morbility and mortality after allogeneic hematopoietic stem cell transplantation (HSCT) with grafts from an HLA-mismatched family donor. Antithymocyteglobulin (ATG) has been widely used to prevent acute GVHD (aGVHD) in haploidentical HSCT. Notwithstanding, immunosuppressive effect of ATG, which may also increase the risk of opportunistic infections, necessitates the use of the lowest possible dose. Till now, the optimal dose of ATG is not known. Here, the investigators compared the outcome of patients receiving haploidentical HSCT treated with two different doses of ATG.

ELIGIBILITY:
Inclusion Criteria:

* Haploidentical hematopoietic stem cell transplant recipient
* Subjects (or their legally acceptable representatives) must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study

Exclusion Criteria:

* Any abnormality in a vital sign (e.g., heart rate, respiratory rate, or blood pressure)
* Patients with any conditions not suitable for the trial (investigators' decision)

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-06; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute GVHD | 1 years
  Acute GVHD was graded according to standard criteria.

SECONDARY OUTCOMES:
Immune reconstitution | 3 years
  Immune reconstitution is performed every 3 months after transplantation.
Survival | 3 years
  Survival includes overall and disease-free survival within 2 years after transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Qifa Liu, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Ottinger HD, Ferencik S, Beelen DW, Lindemann M, Peceny R, Elmaagacli AH, Husing J, Grosse-Wilde H. Hematopoietic stem cell transplantation: contrasting the outcome of transplantations from HLA-identical siblings, partially HLA-mismatched related donors, and HLA-matched unrelated donors. Blood. 2003 Aug 1;102(3):1131-7. doi: 10.1182/blood-2002-09-2866. Epub 2003 Apr 10. PMID 12689945
- [Background] Bacigalupo A, Lamparelli T, Bruzzi P, Guidi S, Alessandrino PE, di Bartolomeo P, Oneto R, Bruno B, Barbanti M, Sacchi N, Van Lint MT, Bosi A. Antithymocyte globulin for graft-versus-host disease prophylaxis in transplants from unrelated donors: 2 randomized studies from Gruppo Italiano Trapianti Midollo Osseo (GITMO). Blood. 2001 Nov 15;98(10):2942-7. doi: 10.1182/blood.v98.10.2942. PMID 11698275